CLINICAL TRIAL: NCT05182047
Title: A Randomized, Open, Crossover, Single Dose, Bioequivalence Study of a Novel Medication Butamirate Citrate Syrup 1.5 mg/mL (McNeil Iberica S.L.U., Spain) vs. Sinecod Syrup (Vanilla) 1.5 mg/mL (GSK Consumer Healthcare S.A., Switzerland), in Adult Healthy Study Volunteers
Brief Title: A Study of Butamirate Citrate Syrup Versus (vs) Sinecod Syrup (Vanilla) in Adult Healthy Study Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision.
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CCSURA001534; CCSURA001534 (Other: McNeil AB)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — butamirate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participant will receive a single oral dose of butamirate citrate syrup 1.5 milligrams per milliliter (mg/mL) (Treatment A [investigational product]) on Day 1 in Treatment Period 1, followed by a single oral dose of sinecod syrup (vanilla) 1.5 mg/mL (Treatment B [Reference product]) on Day 11 in Treatment Period 2. A wash-out period of at least 10 days will be maintained between each treatment period.
  Interventions: Drug: Butamirate citrate; Drug: Sinecod
- Treatment Sequence BA (Experimental): Participants will receive Treatment B on Day 1 in Treatment Period 1, followed by Treatment A on Day 11 in Treatment Period 2. A wash-out period of at least 10 days will be maintained between each treatment period.
  Interventions: Drug: Butamirate citrate; Drug: Sinecod

INTERVENTIONS:
Drug: Butamirate citrate — Butamirate citrate syrup will be administered orally.
Drug: Sinecod — Sinecod syrup will be administered orally.

SUMMARY:
The purpose of this study is to evaluate bioequivalence with respect to rate and extent of absorption of 2-phenylbuturic acid of the novel medication butamirate citrate syrup 1.5 milligrams per milliliter (mg/mL), and the medication sinecod syrup (vanilla) 1.5 mg/mL after single-dose administration in fasting condition by healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female volunteers between the ages of 18 and 45 years, inclusive, with verified diagnosis of healthy: the absence of any gastrointestinal, liver, kidney, cardiovascular, neurologic and infectious or respiratory disease (with no abnormalities as judged by standard clinical, laboratory and instrumental investigations)
* Non- or ex-tobacco users, being defined as someone who completely stopped smoking or using any form of tobacco or nicotine-containing product for at least 12 months before first dose of the study drug in this study
* Volunteers will have a Body Mass Index (BMI) between 18.5 to 30 kilograms per meter square (kg/m^2), inclusive, and a total body weight greater than (>) 50 kg
* For females: Postmenopausal state (absence of menstrual discharge for at least two years and a serum follicle-stimulating hormone [FSH] level exceeding 30 international units per liter [IU/L]) or premenopausal/perimenopausal state with an effective means of contraception (oral, injected, implanted, or transdermal hormonal contraceptives, vaginal contraceptive ring, intrauterine device or status after operative sterilization), during the study and 30 days thereafter, single male partner who has had a vasectomy, or abstinence from heterosexual intercourse during the study and 30 days thereafter
* For males: No pregnant spouse or partner at screening and willingness to utilize an acceptable form of birth control with spouse or any potential partner during the study and 30 days thereafter
* A personally signed and dated informed consent document, indicating that the volunteer has been informed of all pertinent aspects of the study
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol

Exclusion Criteria:

* Hypersensitivity to the ingredients/components of any of the investigational products and/or fructose intolerance
* Burdened history of allergy
* Special diet (that is, vegetarian or vegan diet, salt-restricted diet) or life style (working night shifts, extreme physical exercise)
* Regular (that is, more than once administration) use of any nonprescription or prescription medications other than contraceptives specified in Inclusion criteria #4, within 2 weeks prior to screening
* Use of any nonprescription or prescription medications, profoundly influencing hemodynamics, liver function, Et cetera (etc.) (barbiturates, omeprazole, cimetidine, etc.) within 30 days prior to screening
* Use of any vitamins, dietary and herbal supplements within 14 days prior to screening
* Depot injection or an implant of any drug other than contraceptives specified in Inclusion criteria #4 within 3 months prior to screening
* Females: Confirmed pregnancy or a positive pregnancy test at the screening visit or planning to become pregnant during the duration of the study, and/or breastfeeding
* History of gastrointestinal surgery other than appendectomy
* Cardiovascular, respiratory, neuroendocrine diseases, as well as gastrointestinal, liver, kidney or hematologic disorders
* Positive test for human immunodeficiency virus (HIV) 1 or 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV) or syphilis (WR)
* Acute infectious disease within 4 weeks prior to screening
* Positive nasal or oropharyngeal polymerase chain reaction (PCR) test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) ribonucleic acid (RNA)
* Risk or confirmed SARS-CoV-2 infection (Coronavirus disease 2019 [COVID-19]): a. History of a confirmed or suspected COVID-19 infection in the last 30 days; b. Contact with COVID-19-infected person within 14 days prior to screening or Visit 2; c. Any international travel within 14 days including members in the same household prior to screening or Visit 2; d. Participants with self-reported symptoms within the past 2 weeks prior to screening or Visit 2: i. Unexplained cough, shortness/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, or chest pain/tightness; ii. Body temperature greater than or equal to (>=) 37.5 degree Celsius (°C), measured in axillar area; iii. Or who have used fever or pain reducers within past 2 days of each onsite visit
* Preplanned vaccination within 5 days prior to dosing. (Regarding study visit scheduling: every effort should be made to ensure volunteers receive necessary vaccinations without delay)
* Alcohol consumption that exceeds weekly limits of 10 alcohol units (1 unit is equivalent to 500 milliliters (mL) of beer or 200 mL of wine or 50 mL of spirits) or history of alcoholism
* Consumed alcohol beverage(s) within 48 hours prior to the first scheduled dose of the study drug, positive urine alcohol test at screening, or inability to abstain from alcohol consumption during the entire study period
* History of narcotic substance and/or drug dependence and/or toxicomania and/or drug abuse
* Positive urine screen for narcotic substance abuse
* Use of xanthine containing products (example, coffee, tea, chocolate or cola drink) within 48 hours before each dose of study drug
* Ingestion of food or beverages containing grapefruit, Chinese grapefruit (pomelo) or Seville oranges (including marmalade) within 10 days before the first dose of study drug and throughout the study
* Participation in clinical trials of medicinal products within 90 days prior to screening
* Donation or loss of blood within 3 months prior to the first dose of study drug if the estimated lost blood volume equaled or exceeded 450 mL
* Abnormal results of laboratory and instrumental methods of examinations, including electrocardiogram (ECG) at screening
* Heart rate less than (<) 60 or greater than (>) 90 per minute at rest, or systolic blood pressure <100 or >130 millimeter of mercury (mm Hg), or diastolic blood pressure <70 or >90 mm Hg measured at screening visit
* Preplanned surgery or procedures during the study period, if this may interfere with the conduct of the study
* Any acute or chronic, medical or psychiatric condition(s) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the medically qualified investigator, would make the volunteer inappropriate for entry into this study
* Any psychologic, emotional problems, and any other condition(s) that may interfere with signing of informed consent form or complying with protocol requirements, for example, inability to adequately cooperate with study personnel
* Relationship to persons involved directly with the conduct of the study (that is, principal investigator; sub-investigators; study coordinators; other study personnel; employees or contractors of the sponsor or Johnson & Johnson [J&J] subsidiaries; and the families of each)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-18 (Estimated); Primary Completion 2022-05-05 (Estimated); Study Completion 2022-05-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of 2-phenylbuturic Acid | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose
  Cmax is defined as the maximum observed plasma concentration of 2-phenylbuturic acid.
Area Under the Concentration Versus Time Curve from Start of Drug Administration Until the Time of the Last Measurable 2-phenylbuturic Acid Plasma Concentration (AUC [tau]) | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose
  AUC (tau) is defined as the area under the concentration versus time curve from start of drug administration until the time of the last measurable 2-phenylbuturic acid plasma concentration.

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve Extrapolated to Infinity (AUC [infinity]) of 2-phenylbuturic Acid | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose on Days 1 and 11
  AUC (infinity) is defined as the area under the concentration versus time curve extrapolated to infinity of 2-phenylbuturic acid.
Extrapolated part of Area Under the Concentration Versus Time Curve Extrapolated to Infinity (AUCextrap) of 2-phenylbuturic Acid | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose on Days 1 and 11
  AUCextrap is defined as extrapolated part of AUC (infinity) of 2-phenylbuturic acid.
Time at Which the Maximum Plasma Concentration of 2-phenylbuturic Acid is Observed (Tmax) | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose on Days 1 and 11
  Tmax is defined as the time at which the maximum plasma concentration of 2-phenylbuturic acid is observed.
Terminal Elimination Rate Constant (lambda[z]) for 2-phenylbuturic Acid in Plasma | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose on Days 1 and 11
  Lambda(z) is defined as the rate at which the 2-phenylbuturic acid is removed from the body system.
Terminal Elimination Half-life (t1/2) of 2-phenylbuturic Acid in Plasma | Predose, 0.25, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72 hours postdose on Days 1 and 11
  T1/2 is defined as the time it takes for the 2-phenylbuturic acid plasma concentration to reduce to half of its original value.
Number of Participants With Adverse Events (AEs) | Up to 29 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Number of Participants with AEs by Severity | Up to 29 days
  Number of participants with AEs by severity will be reported. The severity of AEs will be assessed by the medically qualified Investigator or designee using the following general categorical descriptors: a) Mild: awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with the volunteer's usual function or normal everyday activities; b) Moderate: sufficient discomfort is present to cause interference to some extent with the volunteer's usual function or normal everyday activity; c) Severe: extreme distress, causing significant impairment of functioning or incapacitation; interferes significantly with volunteer's usual function; prevents normal everyday activities.
Number of Participants with AE Relationship to Investigational Product Assessment | Up to 29 days
  Number of participants with AE relationship to investigational product assessment will be reported.
Number of Participants with Change from Baseline in Vital Signs Parameters | Up to 29 days
  Number of participants with change from baseline in vital sign parameters (temperature, pulse/heart rate, and blood pressure) will be reported.
Number of Participants with Change from Baseline in Safety Laboratory Parameters | Up to 29 days
  Number of participants with change from baseline in safety laboratory parameters (including physical examination, clinical laboratory tests and electrocardiograms [ECG]) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin A Zakharov, MD, Principal Investigator — "Scientific and Research centre Eco-safety" Limited Liability Company
Locations (1):
- "Scientific and Research centre Eco-safety" Limited Liability Company, 65, Yuri Gagarin prospect, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bohner H, Janiak PS, Nitsche V, Eichinger A, Schutz H. Relative bioavailability of different butamirate citrate preparations after single dose oral administration to 18 healthy volunteers. Int J Clin Pharmacol Ther. 1997 Mar;35(3):117-22. PMID 9089001
- [Background] Faruqi S, Wright C, Thompson R, Morice AH. A randomized placebo controlled trial to evaluate the effects of butamirate and dextromethorphan on capsaicin induced cough in healthy volunteers. Br J Clin Pharmacol. 2014 Dec;78(6):1272-80. doi: 10.1111/bcp.12458. PMID 24995954
- [Background] Miko P. [The use and safety of butamirate containing drops, syrup and depot tablets in Hungary]. Orv Hetil. 2005 Mar 27;146(13):609-12. Hungarian. PMID 15856625
- [Background] Charpin J, Weibel MA. Comparative evaluation of the antitussive activity of butamirate citrate linctus versus clobutinol syrup. Respiration. 1990;57(4):275-9. doi: 10.1159/000195855. PMID 2095610
- [Background] Germouty J, Weibel MA. [Clinical comparison of butamirate citrate with a codeine-based antitussive agent]. Rev Med Suisse Romande. 1990 Nov;110(11):983-6. No abstract available. French. PMID 1980027
- [Background] Lejeune J, Weibel MA. [Comparison of 2 antitussive agents in pediatrics (butamirate citrate in drinkable solution and zipeprol syrup)]. Rev Med Suisse Romande. 1990 Feb;110(2):181-5. No abstract available. French. PMID 2315598
- [Background] Materazzi, F., et al., Note terapeutiche sul butamirato citrato. Gazzetta Medica Italiana - Archivio Scienze Mediche, 1984(143): p. 229-232
- [Background] EMEA Guideline on the Investigation of Bioequivalence, January 2010, CPMP/EWP/QWP/1401/98
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Manual on medicinal products evaluation (in Russian), V.1 (1), 2013. 328 с. FSBI "Scientific Centre for Expert Evaluation of Medicinal Products", Ministry of Health and Family Welfare of the Russian Federation.
- [Background] Resolution # 85 of CEEC "On the Rules for conducting bioequivalence studies of drug products on the territory of EAEU" dated 3-Nov-2016
- [Background] APPENDIX #6 to the "Rules for conducting bioequivalence studies of drug products on the territory of EAEU" dated 3-Nov-2016
- [Background] EMA Guideline on Bioanalytical Method Validation, EMEA/CHMP/EWP/192217/2009
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568